CLINICAL TRIAL: NCT00895765
Title: Part 1 The Outcome of Children With Melamine-Related-Calculus
Brief Title: The Follow up of Chinese Young Children With Melamine-Related-Calculus
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zhejiang University (Other)
Responsible Party: Chao Chun Zou, The Children's Hospital of Zhejiang University
Other Study IDs: zoucc1; 2008ZX007; 20082X010
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Calculus
Keywords: Melamine; Calculus; Kidney; Child
MeSH Terms: conditions — Calculi

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the lesions, clinical features and outcome in young children with melamine-related-calculus.

DETAILED DESCRIPTION:
1. To investigate the outcome of melamine-related-calculus.

   * The change of calculus.
   * The change of obstruction features,including hydronephrosis and ureterectasia.
   * The change of the urinalysis.
2. To investigate the change of renal function in children with melamine-related-calculus during the follow up.

   * Creatinine, urea and uric acid.
   * α and β2 microglobulin.
3. To analysis the factors might be associated with the outcome.

   * The characteristics of patients: age, gender, and so on.
   * The characteristics of calculus: location, size, and so on.

ELIGIBILITY:
Inclusion Criteria:

* children with melamine-related-calculus: with a history of melamine contaminated products
* the parents leave the detailed information for contact and willing to be recalled

Exclusion Criteria:

* children with other congenital renal abnormality
* children with hypercalciuria
* children have abnormality of parathyroid gland

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: young children with melamine-related-calculus
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
The calculus measured by sonography | at 1, 3, 6 and 12 months

SECONDARY OUTCOMES:
Renal function (e.g., creatinine, microglobulin) | at 1, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zou Chao Chun, Master, Principal Investigator — Departemnt of Endocrinology and Children Health care
Locations (1):
- The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China